CLINICAL TRIAL: NCT02546154
Title: A Non-interventional Study of the Time to Relapse of Iron Deficiency Anaemia After Standard Treatment With the Intravenous Iron Monofer® (10% Iron Isomaltoside 1000)
Brief Title: Time to Relapse of Iron Deficiency Anaemia After Standard Treatment With The Intravenous Iron (Monofer®)
Status: Completed | Type: Observational
Sponsor: Pharmacosmos UK Ltd (Industry)
Collaborators: BioStata (Industry)
Responsible Party: Sponsor
Organization: Pharmacosmos A/S (Industry)
Other Study IDs: Monofer-NIS-07
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-03

CONDITIONS: Iron Deficiency Anaemia
Keywords: Iron; Anaemia; Anaemia, Iron-Deficiency; Kidney Diseases; Inflammatory Bowel Diseases; Fatigue
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Kidney Diseases; Inflammatory Bowel Diseases; Fatigue | interventions — iron isomaltoside 1000

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CKD, iron deficiency anaemia: 10% Iron Isomaltoside 1000 administered intravenously to Chronic Kidney Disease patients in doses at the doctor's discretion for treatment of iron deficiency anaemia.
  Interventions: Drug: 10% Iron Isomaltoside 1000
- IBD, iron deficiency anaemia: 10% Iron Isomaltoside 1000 administered intravenously to Inflammatory Bowel Disease patients in doses at the doctor's discretion for treatment of iron deficiency anaemia.
  Interventions: Drug: 10% Iron Isomaltoside 1000

INTERVENTIONS:
Drug: 10% Iron Isomaltoside 1000 — Standard clinical practice and following the Monofer® label (SPC)
  Other Names: Monofer®

SUMMARY:
The objective is to monitor and quality assure the efficacy, including effects on quality of life, and safety of Monofer® in Chronic Kidney Disease and Inflammatory Bowel Disease patient populations when Monofer® is used according to the Monofer® label (Summary of Product Characteristics, SPC) in current clinical practice and where standard routines are being followed.

DETAILED DESCRIPTION:
Intravenous (IV) iron is a well-tolerated and efficacious treatment of iron deficiency anaemia in conditions such as Chronic Kidney Disease (CKD) and Inflammatory Bowel Disease (IBD). Several studies in CKD and IBD patients have shown that IV iron is superior to oral iron, most likely explained by decreased uptake and poor compliance (due to gastrointestinal side-effects) when using oral iron.

The patented Iron Isomaltoside 1000 (Monofer®) has been developed to overcome the current limitations of IV iron drugs with regards to safety and convenience of use. The possibility to administer Monofer® at high single doses (up to 20 mg/kg) reduces the number of treatment visits needed for full iron correction, which is cost-effective, resource and time-sparing, and a reduced drug exposure frequency decreases the risk of side-effects such as infusion reactions.

The objective of the study is to monitor and quality assure the efficacy, including effects on quality of life, and safety of Monofer® in CKD and IBD patient populations when Monofer® is used according to the Monofer® label (Summary of Product Characteristics, SPC) in current clinical practice and where standard routines are being followed. The scientific rationale being to fulfill a need for systematic information/auditing on applied practice including both short and long-term experience with the use of IV iron in different hospital settings and in current clinical practice. The outcome will provide an evidence base for optimised treatment procedures in terms of safety and efficacy.

The total duration of the study per site is approximately 21 months, which includes a 6 months enrollment period, a prospective observation period of at least 12 months, and a period of maximum 3 months prior to the last blood test. Patients will only attend hospital visits planned as part of their standard treatment and they will receive treatment as a part of standard care and according to the doctor's discretion. The number of patient visits depends on the number of Monofer® treatment courses needed during the study period. Each patient can receive one or more treatment courses during 12 months after informed consent. The last blood test will be taken after the last Monofer® treatment course which might occur 13-15 months after informed consent. Study termination will occur once the 12 months observational period has been completed for all patients and the last blood test has been collected from the last Monofer® treated patient in the study. Each treatment course can consist of one or more Monofer® administrations. For each administration of Monofer® either intravenous infusion or injection can be used. Pre- and post-treatment blood tests according to standard treatment and quality of life assessments for fatigue symptoms (FACIT-Fatigue and IBD-F Scales) are a part of the Monofer® treatment course. Laboratory assessments, i.e. anaemia work-up/treatment evaluation, shall be a part of local standard practice. The protocol does not accept any additional samples outside current local standard practice to be taken.

Clinical data management will be performed in accordance with applicable standards and data cleaning procedures. The collected data will systematically be entered into an electronic case report form (eClinicalOS, myEDC, license by BioStata Aps Denmark). The sources of information are the relevant treatment and laboratory results obtained from patient records as well as the quality of life questionnaires for fatigue symptoms. The data will be evaluated by the Pharmacosmos Medical Affairs teams and an external Data Management vendor located in a country within the European Union.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with iron deficiency anaemia as a consequence of CKD or IBD (on the basis of local definition or clinical judgement), treated on the doctor's discretion with Monofer® as standard treatment according to current practice

Exclusion Criteria:

* Patients diagnosed with both CKD and IBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years of age diagnosed with iron deficiency anaemia as a consequence of CKD or IBD.
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Time to relapse of iron deficiency anaemia | From screening until 12 months

SECONDARY OUTCOMES:
Change in scores for fatigue symptoms | Immediately before to earliest 4 weeks after each treatment course during 12 months
Change in anaemia-related blood parameter levels (haemoglobin, iron parameters) | Immediately before to earliest 4 weeks after each treatment course during 12 months
IV iron dose (total needed dose per treatment course) | From screening until 12 months
Number and seriousness of Adverse Drug Reactions | From screening until 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Simon, PhD, Study Chair — Pharmacosmos A/S; Jason Moore, BMedSci, BMBS, FRCP, Principal Investigator — Royal Devon and Exeter Hospital NHS Foundation Trust
Locations (1):
- Royal Devon and Exeter Hospital NHS Foundation Trust, Exeter, United Kingdom

REFERENCES:
- [Derived] Kalra PA, Bhandari S, Spyridon M, Davison R, Lawman S, Mikhail A, Reaich D, Pritchard N, McCafferty K, Moore J. NIMO-CKD-UK: a real-world, observational study of iron isomaltoside in patients with iron deficiency anaemia and chronic kidney disease. BMC Nephrol. 2020 Dec 10;21(1):539. doi: 10.1186/s12882-020-02180-2. PMID 33302891